CLINICAL TRIAL: NCT03045861
Title: A Phase 2a, Multicenter, Randomized, Adaptive, Open-label, Dose Ranging Study to Evaluate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of Cobicistat-boosted GSK2838232 Monotherapy Over 10 Days in HIV-1 Infected Treatment-naive Adults
Brief Title: Safety and Efficacy Study of GSK2838232 in Human Immunodeficiency Virus (HIV)-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200911
Record Dates: First submitted 2017-01-12; First posted 2017-02-08 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — GSK-2838232; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1-GSK2838232 100 mg + Cobicistat 150 mg in Part A (Experimental): During Part A (Cohort 1), subjects will receive a single dose of GSK2838232 100 mg and Cobicistat 150 mg once daily each morning with a light breakfast meal and 240 mL of water from Day 1 to Day 10. Subjects will be followed up to Day 22.
  Interventions: Drug: GSK2838232; Drug: Cobicistat
- Cohort 2-GSK2838232 200 mg + Cobicistat 150 mg in Part B (Experimental): During Part B (Cohort 2), subjects will receive a single dose of GSK2838232 200 mg and Cobicistat 150 mg once daily each morning with a light breakfast meal and 240 mL of water from Day 1 to Day 10. Subjects will be followed up to Day 22.
  Interventions: Drug: GSK2838232; Drug: Cobicistat
- Cohort 3-GSK2838232 50 mg + Cobicistat 150 mg in Part B (Experimental): During Part B (Cohort 3), subjects will receive a single dose of GSK2838232 50 mg and Cobicistat 150 mg once daily each morning with a light breakfast meal and 240 mL of water from Day 1 to Day 10. Subjects will be followed up to Day 22.
  Interventions: Drug: GSK2838232; Drug: Cobicistat
- Cohort 4-GSK2838232 20 mg + Cobicistat 150 mg in Part B (Experimental): During Part B (Cohort 4), subjects will receive a single dose of GSK2838232 20 mg and Cobicistat 150 mg once daily each morning with a light breakfast meal and 240 mL of water from Day 1 to Day 10. Subjects will be followed up to Day 22.
  Interventions: Drug: GSK2838232; Drug: Cobicistat

INTERVENTIONS:
Drug: GSK2838232 — GSK2838232 capsules will be supplied as swedish orange, unmarked capsule (50 mg), and white, unmarked capsules (10 mg) in high-density polyethylene bottles.
Drug: Cobicistat — Cobicistat tablets 150 mg will be supplied as an orange, round, biconvex, film-coated tablet in bulk containers for individualized dosing.

SUMMARY:
GSK2838232 is a novel HIV-1 maturation inhibitor (MI) that is being developed for the treatment of HIV-1 infection in combination with other antiretroviral therapy (ART). This study will be a 10-day monotherapy, open-label, adaptive, dose ranging, repeat-dose study. This study will be conducted in two Parts (Part A and Part B) consisting single daily doses of GSK2838232 and Cobicistat from Day 1 to Day 10. This proof of concept open-label study will be aimed to characterize the acute antiviral activity, pharmacokinetics (PK), the relationship between PK and antiviral activity, and safety of GSK2838232/cobi administered across a range of doses over 10 days in HIV-1 infected patients. A cohort of 10 subjects will be studied in Part I followed by interim (go/no-go) analysis of Part A data. On completion of an interim analysis of part A data, further cohorts of 8 subjects will then be studied in Part B in a parallel design in two or more cohorts (depending upon the data obtained in Part A). Approximately 34 HIV-1 infected treatment-naive subjects will be enrolled during the study. Subjects in both parts will have a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose. Maximum duration of study participation will be approximately 6 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy (other than HIV infection) male or female as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring, defined as no other chronic medical conditions and taking no chronic medications.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the medical monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A creatinine clearance >80 mL/minute as determined by Cockcroft-Gault equation creatinine clearance CLcr (mL/minute) = (140 - age) x weight (Wt) divided by (72 x serum creatinine [Scr]) (times 0.85 if female) where age is in years, Wt is in kilogram (kg), and Scr is in units of mg/decilitre (dL).
* Confirmed HIV positive; CD4+ cell count >=350 cells/millimetre (mm)^3 and plasma HIV-1 RNA >=5000 copies/mL at screening.
* No current and no prior ART.
* Body weight >=50 kg (110 pound [lbs.]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/meter^2 (inclusive)
* A female subject of reproductive or non-reproductive potential is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin (hCG) test at screening and prior to first dose), not lactating, and at least one of the following conditions applies: females of reproductive potential may only be enrolled if they are using two forms of complementary contraception, which must include one barrier method. They will be counselled on safer sex practices; there is no definitive drug-drug interaction (DDI) information with GSK2838232 and an interaction with oral contraceptives is possible, so other (barrier, inter-uterine device etc.) methods of contraception will be required; fertile females, who have an established, long-term lifestyle of sexual abstinence, or only same sex partners, require no other means of birth control. Pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented bilateral oophorectomy; postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until one week after the last dose of study medication; vasectomy with documentation of azoospermia; male condom plus partner use of one of the contraceptive options as: Contraceptive sub dermal implant including a <1 percent rate of failure per year; intrauterine device or intrauterine system including a <1 percent rate of failure per year; oral contraceptive, either combined or progestogen alone or injectable progestogen; contraceptive vaginal ring; percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin (BIL) >1.5 x upper limit of normal (ULN), isolated BIL >1.5xULN is acceptable if BIL is fractionated and direct BIL <35 percent.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); hepatitis B virus (HBV) and/or hepatitis C virus (HCV) positive.
* Subjects who have any other chronic medical condition, including cardiovascular (CV), respiratory, neurologic, psychiatric, renal, gastrointestinal (GI), oncologic, rheumatologic, or dermatologic.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Smoking is an exclusion criteria for this study. Subject having urinary cotinine levels indicative of smoking at screening.
* Chronic marijuana or use of other elicit medications (cocaine, heroin) is an exclusion criteria.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Screening or Baseline cardiac troponin I greater than the 99 percent cutoff (>0.045 nanogram [ng]/mL by the Dimension Vista cardiac troponin [CTN] I assay).
* A positive pre-study drug/alcohol screen.
* Prior history of receiving an HIV maturation inhibitor
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of study drug administration or anticipated need for such treatment within the study.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration.
* An active Center for Disease Control and Prevention (CDC) category C disease except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.
* Treatment with any vaccine within 30 days prior to receiving study medication.
* Exclusion criteria for 24-hour screening holter: any symptomatic arrhythmia (except isolated extra systoles); sustained cardiac arrhythmias (such as atrial fibrillation, flutter or supraventricular tachycardia [>=10 seconds]); non-sustained or sustained ventricular tachycardia (defined as >=3 consecutive ventricular ectopic beats); any conduction abnormality including but not specific to left or complete bundle branch block, atrioventricular (AV) block, high grade or complete heart block Wolff-Parkinson-White (WPW) syndrome etc.; sinus pauses >3 seconds.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): heart rate <45 and >100 beats per minute (bpm) for males, and <50 and >100 bpm for females; PR Interval <120 and >220 milliseconds (msec); QRS duration <70 and >120 msec; corrected QT (QTc) interval >450 msec; Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization); any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome); sinus pauses >3 seconds; any significant arrhythmia which, in the opinion of the principal investigator or GSK medical monitor, will interfere with the safety for the individual subject; non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (11):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Longview, Texas
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20281

REFERENCES:
- [Background] DeJesus E, Harward S, Jewell RC, Johnson M, Dumont E, Wilches V, Halliday F, Talarico CL, Jeffrey J, Gan J, Xu J, Felizarta F, Scribner A, Ramgopal M, Benson P, Johns BA. A Phase IIa Study Evaluating Safety, Pharmacokinetics, and Antiviral Activity of GSK2838232, a Novel, Second-generation Maturation Inhibitor, in Participants With Human Immunodeficiency Virus Type 1 Infection. Clin Infect Dis. 2020 Aug 22;71(5):1255-1262. doi: 10.1093/cid/ciz938. PMID 31769793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a dose ranging study to evaluate the antiviral effect, safety, tolerability and pharmacokinetics of cobicistat-boosted GSK2838232 monotherapy over 10 days in human immunodeficiency virus-1 (HIV-1) infected participants.
Pre-assignment Details: A total of 85 participants were screened across 21 sites in the United States and Canada of which 52 participants failed screening. Thirty three participants were enrolled from 15 sites in the United States and Canada.
Groups:
- GSK2838232 20 mg: Eligible HIV-1 infected participants were administered a single oral dose of GSK2838232 20 milligrams (mg) and 150 mg cobicistat once daily with a light breakfast meal and 240 milliliters (mL) of water from Day 1 to Day 10.
- GSK2838232 50 mg: Eligible HIV-1 infected participants were administered a single oral dose of GSK2838232 50 mg and 150 mg cobicistat once daily with a light breakfast meal and 240 mL of water from Day 1 to Day 10.
- GSK2838232 100 mg: Eligible HIV-1 infected participants were administered a single oral dose of GSK2838232 100 mg and 150 mg cobicistat once daily with a light breakfast meal and 240 mL of water from Day 1 to Day 10.
- GSK2838232 200 mg: Eligible HIV-1 infected participants were administered a single oral dose of GSK2838232 200 mg and 150 mg cobicistat once daily with a light breakfast meal and 240 mL of water from Day 1 to Day 10.
Period: Part A (Up to 10 Days)
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Started | 0 | 0 | 10 | 0
Completed | 0 | 0 | 10 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part B (Up to 10 Days)
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Started | 7 | 8 | 0 | 8
Completed | 7 | 8 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg | Total
Number analyzed (Participants) | 7 | 8 | 10 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (5.59) | 25.4 (9.74) | 31.8 (10.66) | 35.8 (14.87) | 29.8 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1
  Male | 7 | 8 | 9 | 8 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, customized: American Indian or Alaska native | 1 | 0 | 1 | 0 | 2
  Race, customized: Asian-South East Asian Heritage | 1 | 0 | 0 | 0 | 1
  Race, customized: Black or African American | 0 | 1 | 5 | 2 | 8
  Race, customized: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Race, customized: White-White/Caucasian/European Heritage | 5 | 6 | 4 | 5 | 20
  Race, customized: Multiple-Black or African American and White | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Decline From Baseline in Plasma HIV-1 Ribonucleic Acid (RNA)
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. An HIV-1 RNA polymerase chain reaction (PCR) assay with a lower limit of detection (LLOD) of 50 copies/milliliter (ultrasensitive assay) was used for post-baseline assessments. Baseline value was the value at latest pre-dose assessment. The maximum decline was determined using change from Baseline in plasma HIV-RNA values at each time point. The analysis was performed on Intent To Treat (ITT) Population which comprised of all participants who met study criteria and were enrolled into the study with documented evidence of having received at least 1 dose of treatment and at least one post-Baseline HIV-1 RNA measurement.
Time Frame: Baseline (Day 1) to Day 21
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Copies per milliliter | -42095.14 (37575.520) | -49065.88 (71339.743) | -32947.50 (54291.492) | -33149.13 (31785.663)

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other important medical events; is associated with liver injury and impaired liver function. Safety Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  Any AEs | 3 | 3 | 5 | 5
  Any SAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: carbon dioxide/bicarbonate (low: <18 millimoles per liter [mmol/L] and high: >32 mmol/L); urea (high: >9 mmol/L); creatinine (high: change from Baseline >44.2 micromoles per liter [µmol/L]), glucose (low: <3 and high: >9 mmol/L); potassium (low: <3 and high: >5.5 mmol/L); troponin I (high: >=0.01 micrograms per liter [µg/L]) and sodium (low: <130 mmol/L and high: >150 mmol/L). Data for any visit post-Baseline is reported.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  Carbon dioxide/bicarbonate; >32 mmol/L | 0 | 0 | 0 | 0
  Carbon dioxide/bicarbonate; <18 mmol/L | 0 | 0 | 3 | 0
  Urea; >9 mmol/L | 1 | 0 | 0 | 0
  Creatinine; Change >44.2 mmol/L | 0 | 0 | 0 | 0
  Glucose; >9 mmol/L | 0 | 0 | 0 | 0
  Glucose; <3 mmol/L | 0 | 0 | 0 | 0
  Potassium; >5.5 mmol/L | 0 | 0 | 0 | 2
  Potassium; <3 mmol/L | 0 | 0 | 0 | 0
  Sodium; >150 mmol/L | 0 | 0 | 0 | 0
  Sodium; <130 mmol/L | 0 | 0 | 0 | 0
  Troponin I; >=0.01 µg/L | 7 | 8 | 10 | 8

4. Primary Outcome: Number of Participants With Hematology Parameter Abnormalities of Potential Clinical Importance
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood); hemoglobin (high: >180 grams per liter [g/L]), lymphocytes (low: <0.8x10^9 cells/L); neutrophil count (low: <1.5x10^9 cells/L); platelet count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); white blood cells (low: <3x10^9 cells/L and high: >20x10^9cells/L). Data for any visit post-Baseline is reported.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  Hematocrit; >0.54 | 0 | 0 | 1 | 1
  Hematocrit; decline from Baseline >0.075 | 1 | 1 | 3 | 0
  Hemoglobin; >180 | 0 | 0 | 0 | 0
  Hemoglobin; decline from Baseline >25 | 0 | 0 | 1 | 0
  Lymphocytes; <0.8 | 0 | 0 | 0 | 0
  Neutrophils; <1.5 | 1 | 0 | 3 | 1
  Platelets; >550 | 0 | 0 | 0 | 0
  Platelets; <100 | 0 | 0 | 1 | 0
  White blood cells; >20 | 0 | 0 | 0 | 0
  White blood cells; <3 | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Liver Function Laboratory Abnormalities of Potential Clinical Importance
Description: Blood samples were collected for the assessment of liver function parameters. The clinical concern range for liver function parameters were: albumin (low: <30 g/L), total protein (low: <15 and high: >15 g/L), alanine aminotransferase (high: >=2 times upper limit of normal [ULN]); aspartate aminotransferase (high: >=2 times ULN); alkaline phosphatase (high: >=2 times ULN); total bilirubin (high: >=1.5 times ULN); direct bilirubin (high: >0.3 times ULN).
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  Albumin; <30 | 0 | 0 | 0 | 0
  Total Protein; ULN+15 | 0 | 0 | 0 | 0
  Total Protein; lower limit of normal (LLN)-15 | 0 | 0 | 0 | 0
  ALT; >=2 times ULN | 0 | 0 | 0 | 0
  AST; >=2 times ULN | 0 | 1 | 0 | 0
  ALP; >=2 times ULN | 0 | 0 | 0 | 0
  Total bilirubin; >=1.5 times ULN | 0 | 0 | 1 | 0
  Direct bilirubin; >=0.3 times ULN | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Urine Parameters
Description: Urine samples were collected for the assessment of following urine parameters by dipstick method: pH, glucose, protein, blood and ketones. The number of participants with abnormal urine parameters is presented.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals. Number of participants with abnormal ECG findings at worst-case post Baseline is presented.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  Abnormal-not clinically significant | 5 | 6 | 8 | 4
  Abnormal-clinically significant | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Vital Signs Data Outside Clinical Concern Range
Description: Vital signs were measured in a semi-supine position after 5 minutes rest and included temperature, systolic and diastolic blood pressure and pulse rate. The clinical concern range for vital signs were: systolic blood pressure (SBP) (low: <85 and high: >160 millimeters of mercury [mmHg]) and diastolic blood pressure (DBP) (low: <45 and high: >100 mmHg). Number of participants with vital signs data outside clinical concern range is presented.
Time Frame: Day 1 (pre-dose)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  SBP; >Clinical concern range | 0 | 0 | 1 | 0
  SBP; <Clinical concern range | 0 | 0 | 0 | 0
  DBP; >Clinical concern range | 0 | 0 | 1 | 0
  DBP; <Clinical concern range | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants Who Were Administered Concomitant Medications
Description: Concomitant medications (prescription and non-prescription) were administered only as medically necessary during the study. Number of participants who received any concomitant medications is presented.
Time Frame: Up to Day 22
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants | 2 | 3 | 3 | 3

10. Primary Outcome: Area Under the Plasma Concentration Time Curve From Zero (Pre-dose) to 24 Hours (AUC[0 to 24]) for GSK2838232 on Day 1
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232. The analysis was performed on Pharmacokinetic Population which comprised of participants who received GSK2838232 and underwent plasma pharmacokinetic sampling during the study.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: Pharmacokinetic Population. One participant from GSK2838232 100 mg arm was dosed with GSK2838232 50 mg on Days 1 and 2; hence, pharmacokinetic parameters for that participant were summarized with GSK2838232 50 mg for Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 9 | 8
Hours*nanograms per milliliter | 187 (35.5) | 453 (60.4) | 966 (67.4) | 2752 (51.7)

11. Primary Outcome: Maximum Observed Concentration (Cmax) for GSK2838232 on Day 1
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 9 | 8
Nanograms per milliliter | 12.65 (36.4) | 32.39 (61.0) | 65.62 (76.7) | 190.0 (44.3)

12. Primary Outcome: Time to Maximum Observed Concentration (Tmax) for GSK2838232 on Day 1
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 9 | 8
Hours | 4.033 [3.00 to 8.00] | 3.250 [2.00 to 8.00] | 6.000 [3.00 to 8.00] | 4.000 [2.00 to 6.00]

13. Primary Outcome: Absorption Lag Time (Tlag) for GSK2838232 on Day 1
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 9 | 8
Hours | 1.083 [0.50 to 1.58] | 1.000 [0.00 to 1.53] | 0.500 [0.00 to 1.50] | 0.500 [0.00 to 1.00]

14. Primary Outcome: Concentration of GSK2838232 at 24 Hours Post-dose on Day 1
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: 24 hours post-dose on Day 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 9 | 8
Nanograms per milliliter | 5.890 (27.6) | 13.45 (87.3) | 30.72 (58.3) | 87.33 (54.6)

15. Primary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC [0 to Tau]) for GSK2838232 on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Hours*nanograms per milliliter | 590 (33.4) | 1024 (40.8) | 2727 (53.1) | 5664 (67.1)

16. Primary Outcome: Pre-dose Concentration (C0) of GSK2838232 on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Nanograms per milliliter | 20.02 (28.8) | 36.66 (39.8) | 75.31 (57.0) | 155.5 (64.5)

17. Primary Outcome: Concentration at End of Dosing Interval (Ctau) for GSK2838232 on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Nanograms per milliliter | 19.24 (33.7) | 31.76 (53.8) | 78.98 (58.3) | 180.3 (79.8)

18. Primary Outcome: Cmax for GSK2838232 on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Nanograms per milliliter | 32.65 (30.8) | 56.40 (33.0) | 157.9 (54.0) | 306.5 (59.2)

19. Primary Outcome: Apparent Oral Clearance of GSK2838232 Following Administration on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Liters per hour | 33.91 (33.4) | 48.84 (40.8) | 36.67 (53.1) | 35.31 (67.1)

20. Primary Outcome: Terminal Elimination Half-life (T1/2) of GSK2838232 Following Administration on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 4 | 5 | 10 | 7
Hours | 19.221 (17.1) | 16.298 (24.0) | 18.113 (18.3) | 16.351 (8.8)

21. Primary Outcome: Tmax for GSK2838232 Following Administration on Day 10
Description: Serial plasma samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232.
Time Frame: Pre dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time point were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Hours | 6.000 [4.00 to 8.00] | 4.000 [2.00 to 8.05] | 6.000 [3.00 to 8.10] | 4.083 [2.00 to 6.00]

22. Secondary Outcome: Change From Baseline to Day 11 in log10 Plasma HIV-1 RNA Relative to Day 10 AUC (0 to Tau)
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Change from Baseline is the value at indicated time point minus Baseline value. Statistical analysis for relationship between pharmacokinetic parameters (AUC) and pharmacodynamic measures (Change from Baseline in plasma HIV-1 RNA) was explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: maximum response (Emax), pharmacokinetic parameter value that attains 50% of the maximal effect (ED50) and residual variability (s2e). Pharmacokinetic/Pharmacodynamic Population comprised of participants who met criteria for Per-Protocol (all participants who met study criteria and are enrolled into the study with documented evidence of having received all doses and all post-baseline HIV-1 RNA measurement, with exceptions of those who have at least one major protocol deviation) and Pharmacokinetic Population analysis sets and who underwent pharmacodynamic sampling during study.
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 8
log10 copies per milliliter | -0.4979 (0.44873) | -1.1671 (0.51996) | -1.1745 (0.45005) | -1.5994 (0.32718)
Statistical Analysis 1: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; Emax = -1.822, 95% CI 2-sided [-2.333 to 1.310]
Statistical Analysis 2: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; ED50 = 1020.755, 95% CI 2-sided [100.786 to 1940.724]
Statistical Analysis 3: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; s2e = 0.200, 95% CI 2-sided [0.095 to 0.306]

23. Secondary Outcome: Change From Baseline to Day 11 in log10 Plasma HIV-1 RNA Relative to Day 10 Cmax
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Change from Baseline is the value at indicated time point minus Baseline value. Statistical analysis for the relationship between pharmacokinetic parameters (Cmax) and pharmacodynamic measures (change from Baseline in log10 plasma HIV-1 RNA) was explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: maximum response (Emax), pharmacokinetic parameter value that attains the 50% of the maximal effect (ED50) and s2e.
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 8
log10 copies per milliliter | -0.4979 (0.44873) | -1.1671 (0.51996) | -1.1745 (0.45005) | -1.5994 (0.32718)
Statistical Analysis 1: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; Emax = -1.801, 95% CI 2-sided [-2.319 to -1.283]
Statistical Analysis 2: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; ED50 = 55.572, 95% CI 2-sided [3.565 to 107.579]
Statistical Analysis 3: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; s2e = 0.206, 95% CI 2-sided [0.097 to 0.314]

24. Secondary Outcome: Change From Baseline to Day 11 in log10 Plasma HIV-1 RNA Relative to Day 10 Ctau
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Change from Baseline is the value at indicated time point minus Baseline value. Statistical analysis for the relationship between pharmacokinetic parameters (Ctau) and pharmacodynamic measures (change from Baseline in log10 plasma HIV-1 RNA) was explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: maximum response (Emax), pharmacokinetic parameter value that attains the 50% of the maximal effect (ED50) and s2e.
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 8
log10 copies per milliliter | -0.4979 (0.44873) | -1.1671 (0.51996) | -1.1745 (0.45005) | -1.5994 (0.32718)
Statistical Analysis 1: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; Emax = -1.846, 95% CI 2-sided [-2.352 to -1.340]
Statistical Analysis 2: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; ED50 = 32.415, 95% CI 2-sided [4.687 to 60.143]
Statistical Analysis 3: Comparison: GSK2838232 20 mg vs GSK2838232 50 mg vs GSK2838232 100 mg vs GSK2838232 200 mg; Test type: Other; s2e = 0.200, 95% CI 2-sided [0.094 to 0.305]

25. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Count to Day 11
Description: CD4+ cell counts were assessed by flow cytometry. Baseline value is the latest pre-dose assessment value. Change from Baseline is calculated as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Day 11
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 8
Cells per microliter | -1.4 (95.26) | 52.0 (145.36) | 40.7 (94.47) | 11.1 (75.15)

26. Secondary Outcome: Change From Baseline to Day 11 in CD4+ Count Relative to Day 10 AUC (0 to Tau)
Description: The relationship between pharmacokinetic parameters (AUC) and pharmacodynamic measures (change from Baseline CD4+ cell count) was explored using a frequentist linear model. The model parameters estimated included slope and intercept. The estimate (slope) along with 95% confidence interval is presented.
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population
Measure: Number (95% Confidence Interval); unit: cells/microliter/ng*h/mL
Groups:
- Participants Receiving GSK2838232: Participants who received GSK2838232 at doses of 20 mg, 50 mg, 100 mg and 200 mg were included.
Arm/Group | Participants Receiving GSK2838232
Number analyzed (Participants) | 31
cells/microliter/ng*h/mL | -0.003 [-0.016 to 0.010]

27. Secondary Outcome: Change From Baseline to Day 11 in CD4+ Count Relative to Day 10 Cmax
Description: The relationship between pharmacokinetic parameters (Cmax) and pharmacodynamic measures (change from Baseline CD4+ cell count) was explored using a frequentist linear model. The model parameters estimated included slope and intercept. The estimate (slope) along with 95% confidence interval is presented
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population
Measure: Number (95% Confidence Interval); unit: cells/microliter/nanograms/milliliter
Arm/Group | Participants Receiving GSK2838232
Number analyzed (Participants) | 31
cells/microliter/nanograms/milliliter | -0.067 [-0.320 to 0.187]

28. Secondary Outcome: Change From Baseline to Day 11 in CD4+ Count Relative to Day 10 Ctau
Description: The relationship between pharmacokinetic parameters (Ctau) and pharmacodynamic measures (change from Baseline CD4+ cell count) was explored using a frequentist linear model. The model parameters estimated included slope and intercept. The estimate (slope) along with 95% confidence interval is presented.
Time Frame: Baseline (Day 1), Days 10 and 11
Population: Pharmacokinetic/Pharmacodynamic Population
Measure: Number (95% Confidence Interval); unit: cells/microliter/nanograms/milliliter
Arm/Group | Participants Receiving GSK2838232
Number analyzed (Participants) | 31
cells/microliter/nanograms/milliliter | -0.079 [-0.451 to 0.292]

29. Secondary Outcome: Number of Participants With Emergent Drug Resistance Mutations
Description: Plasma samples were collected to evaluate treatment-emergent genotypic mutations in Gag, reverse transcriptase (RT) and protease (PR) and to assess phenotypic resistance to GSK2838232 and RT and PR drugs. Number of participants with treatment emergent RT/PR mutations, reduced susceptibility to nucleoside/nucleotide reverse transcriptase inhibitor (NRTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), or protease inhibitor (PI), treatment emergent maturation inhibitor A364A/V and GSK2838232 phenotypic resistance is presented.
Time Frame: Up to Day 11
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Participants
  RT/PR mutations | 0 | 0 | 0 | 0
  Reduced susceptibility to NRTIs, NNRTIs, PIs | 0 | 0 | 0 | 0
  GSK2838232 phenotypic resistance | 0 | 1 | 0 | 0
  Treatment emergent A364A/V | 0 | 1 | 1 | 0

30. Secondary Outcome: Accumulation Ratio for GSK2838232
Description: Serial blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232. The accumulation ratios were calculated as R_AUC=AUC(0-tau) Day 10/AUC(0-24) Day 1; R_Cmax=Cmax Day 10/Cmax Day 1 and R_Ctau=Ctau Day 10/C24 Day 1.
Time Frame: pre dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Days 1 and 10; pre-dose on Days 3, 4, 5, 8 and 9; Days 12 and 14
Population: Pharmacokinetic Population. Only participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 7 | 10 | 7
Ratio
  R_AUC | 3.149 (42.2) | 2.004 (34.4) | 3.229 (46.1) | 2.211 (27.2)
  R_Cmax | 2.580 (45.1) | 1.498 (40.0) | 2.753 (43.4) | 1.668 (26.5)
  R_Ctau | 3.267 (41.2) | 2.118 (43.9) | 3.038 (64.8) | 2.210 (45.1)

31. Secondary Outcome: Dose Proportionality of GSK2838232
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232. Dose proportionality was assessed using a fixed effects power model. Estimated slope and 90% confidence interval is presented.
Time Frame: pre dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Days 1 and 10
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category )
Measure: Number (90% Confidence Interval); unit: slope of log dose
Arm/Group | Participants Receiving GSK2838232
Number analyzed (Participants) | 33
slope of log dose
  AUC(0-24); Day 1 | 1.157 [0.971 to 1.343]
  Cmax; Day 1 | 1.158 [0.968 to 1.349]
  C24; Day 1 | 1.170 [0.968 to 1.371]
  AUC (0 to tau); Day 10 | 1.012 [0.835 to 1.190]
  Cmax; Day 10 | 1.013 [0.845 to 1.181]
  Ctau; Day 10 | 0.988 [0.787 to 1.190]

32. Secondary Outcome: Pre-morning Dose Concentrations (C0) on Day 2 Through 11
Description: Blood samples were collected for pharmacokinetic analysis of GSK2838232. The pre-morning dose concentrations for Days 2 to 11 is presented. One participant from GSK2838232 100 mg arm was dosed with GSK2838232 50 mg on Days 1 and 2; hence, pharmacokinetic parameters for that participant were summarized with GSK2838232 50 mg for Days 1 and 2 and with GSK2838232 100 mg for Days 3 to 10.
Time Frame: Pre-dose on Days 2, 3, 4, 5, 8, 9, 10 and 11
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 9 | 10 | 8
Nanograms per milliliter
  Day 2; n=7, 9, 9, 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Day 2; n=7, 9, 9, 8 | 6.08 (1.695) | 16.39 (9.002) | 34.17 (13.990) | 96.94 (44.319)
  Day 3; n=7, 8, 10, 8: number analyzed (Participants) | 7 | 8 | 10 | 8
  Day 3; n=7, 8, 10, 8 | 13.99 (5.576) | 29.03 (11.870) | 51.27 (25.971) | 163.98 (91.368)
  Day 4; n=7, 7, 10, 8: number analyzed (Participants) | 7 | 7 | 10 | 8
  Day 4; n=7, 7, 10, 8 | 14.66 (5.771) | 31.80 (13.319) | 64.49 (26.710) | 176.28 (96.684)
  Day 5; n=4, 6, 10, 7: number analyzed (Participants) | 4 | 6 | 10 | 7
  Day 5; n=4, 6, 10, 7 | 15.03 (3.308) | 34.35 (15.626) | 76.14 (35.179) | 206.29 (69.533)
  Day 8; n=7, 8, 10, 8: number analyzed (Participants) | 7 | 8 | 10 | 8
  Day 8; n=7, 8, 10, 8 | 19.72 (7.139) | 43.14 (16.664) | 86.39 (43.382) | 187.16 (110.304)
  Day 9; n=7, 6, 10, 8: number analyzed (Participants) | 7 | 6 | 10 | 8
  Day 9; n=7, 6, 10, 8 | 20.53 (6.760) | 43.83 (18.691) | 89.32 (40.407) | 206.75 (124.166)
  Day 10; n=7, 7, 10, 8: number analyzed (Participants) | 7 | 7 | 10 | 8
  Day 10; n=7, 7, 10, 8 | 20.76 (6.426) | 39.19 (16.502) | 84.52 (39.940) | 189.05 (107.636)
  Day 11; n=7, 7, 10, 8: number analyzed (Participants) | 7 | 7 | 10 | 8
  Day 11; n=7, 7, 10, 8 | 20.16 (6.828) | 35.09 (16.038) | 89.87 (49.195) | 219.23 (133.552)

33. Secondary Outcome: Steady State Assessment of Plasma Pre-dose Concentrations by Treatment
Description: A linear mixed model using Day, treatment and Day by treatment as fixed effects and participant as a random effect on the log-transformed pre-dose values was performed to evaluate if steady state was achieved using the Helmert transformation approach. The comparison was done as Day 8 versus the average of Days 9 and 10 values. The ratio of geometric least square mean for Day 8 versus average of Days 9 and 10 values is presented along with 95% confidence interval.
Time Frame: Pre-dose on Days 8, 9 and 10
Population: Pharmacokinetic Population
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
Number analyzed (Participants) | 7 | 8 | 10 | 8
Ratio | 0.924 [0.778 to 1.097] | 0.999 [0.839 to 1.189] | 0.958 [0.830 to 1.106] | 0.961 [0.818 to 1.128]

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from the start of study treatment until Day 22
Description: SAEs and non-serious AEs were collected in the Safety Population
Arm/Group | GSK2838232 20 mg | GSK2838232 50 mg | GSK2838232 100 mg | GSK2838232 200 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 3/7 | 3/8 | 5/10 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2838232 20 mg (N=7) | GSK2838232 50 mg (N=8) | GSK2838232 100 mg (N=10) | GSK2838232 200 mg (N=8)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03045861/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03045861/SAP_001.pdf